CLINICAL TRIAL: NCT03276390
Title: A Culturally Targeted Transplant Program to Increase Live Donation in Hispanics
Brief Title: A Culturally Targeted Transplant Program
Acronym: HKTP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Mayo Clinic (Other); Baylor Health Care System (Other); University of Colorado, Denver (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Elisa Gordon, Professor, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01DK104876-01 (NIH)
Record Dates: First submitted 2017-09-05; First posted 2017-09-08 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: ESRD
Keywords: health disparities; living donation
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Two group comparison (intervention vs. control) and pre-post comparison (within each site).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention study site (Active Comparator): Exposure to the intervention, which is the Northwestern Medicine (TM) Hispanic Kidney Transplant Program, a culturally targeted program for Hispanic potential recipients for transplant evaluation that is implemented into the 2 study sites.
  The intervention study site will provide the intervention to its Hispanic patients.
  The intervention study will will also provide the routine care (control arm) to all other patients.
  For the purposes of this study, Hispanic potential recipients recruited into the study will be exposed to this intervention. Non-Hispanic Whites recruited into the study will not be exposed to this intervention.
  Interventions: Behavioral: Hispanic Kidney Transplant Program (HKTP)
- No intervention study site (No Intervention): Exposure to routine transplant evaluation at the two control sites.

INTERVENTIONS:
Behavioral: Hispanic Kidney Transplant Program (HKTP) — The HKTP entails culturally targeted education in Spanish about transplantation, outreach to dialysis patients by bicultural health care providers.
  Arms: Intervention study site

SUMMARY:
Hispanic/Latino patients with end-stage renal disease are disproportionately less likely to get a kidney transplant, and specifically, a living donor kidney transplant (LDKT), compared to non-Hispanic whites. Accordingly, without LDKTs, Hispanics experience longer transplant waiting times, shorter patient and graft survival, and worse quality of life. Cultural beliefs and linguistic barriers contribute to the disparity in LDKTs. The objective of the proposed study is to implement and evaluate Northwestern Medicine's® Hispanic Kidney Transplant Program, a culturally-competent transplant center-based intervention, at two transplant centers serving large Hispanic populations. The proposed study will provide valuable knowledge about the potential to rapidly disseminate the HKTP as a novel approach to increase Hispanic LDKTs nationally.

DETAILED DESCRIPTION:
The shortage of organs for kidney transplantation for patients with end-stage renal disease (ESRD) is magnified in Hispanics/Latin Americans. Hispanics have a disproportionately higher prevalence of ESRD, yet receive fewer kidney transplants compared to non-Hispanic whites. Living donor kidney transplant (LDKT) is the treatment of choice for ESRD as it confers better patient and graft survival, shorter waiting time, and better quality of life than deceased donor kidney transplantation. However, compared to their representation on the waiting list, fewer Hispanics received a LDKT than non-Hispanic whites in 2013: 4% versus 10%. Barriers to LDKT for Hispanics include: lack of knowledge, cultural concerns, and language barriers. The disparity will likely worsen without intervention as Hispanics are the largest and fastest growing minority group in the US.

Few available culturally competent interventions have led to increased LDKT rates. Interventions rarely address Hispanic cultural concerns, and there are no published models of transplant center-based only programs. The Chicago Northwestern Medicine's® Hispanic Kidney Transplant Program (HKTP), a culturally and linguistically competent program, has increased Hispanic LDKTs. The mean annual ratio of Hispanic to non-Hispanic white LDKTs grew from 0.20 in 2001-2006 to 0.34 in 2008-2013, a 70% increase (p<0.001).

The objective of this study is to implement and evaluate the HKTP, a culturally-competent transplant center-based intervention, at two transplant centers serving large Hispanic populations (Dallas, TX, and Los Angeles, CA), with Northwestern University serving as the Study Coordinating Center. The pre-post HKTP intervention study will evaluate the effect of the HKTP's key culturally sensitive components (outreach, communication, education) on Hispanic LDKT rates, compared to matched controls. The specific aims are to:

1. Implement the HKTP at two transplant centers by conducting a needs assessment of barriers and using a "learning collaborative" model to deliver HKTP protocols, scripts, and materials.
2. Conduct a pre-post HKTP intervention evaluation with matched controls to assess if the HKTP is associated with an increase in: a) the ratio of Hispanic to non-Hispanic white LDKTs as a function of an absolute increase in Hispanic LDKTs, b) ESRD Hispanic patient additions to the waiting list, c) Hispanic potential donors per potential recipient, and d) Hispanic patients' satisfaction with care.
3. Formatively evaluate the fidelity and innovative adaptations to HKTP's outreach, communication, and education at both study sites to identify effective components of the HTKP, using mixed methods.

As an exploratory aim, a budget impact analysis will be conducted to construct a business case for transplant centers and permit estimates of HKTP scalability. The proposed study will provide valuable knowledge about the potential to rapidly disseminate the HKTP as a novel approach to increase Hispanic LDKTs nationally, improve health outcomes for Hispanics, and close the LDKT disparity gap.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic or non-Hispanic white potential recipients initiating evaluation for a transplant
* age 18 or older
* The above potential recipients' potential donors initiating evaluation for living donation

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11836 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Ratio of Hispanic to non-Hispanic white LDKTs | Post-intervention exposure up to 3.5 years
  A center-level variable. This is a metric of disparity

SECONDARY OUTCOMES:
Number of Hispanic living kidney donors | Post-intervention exposure up to 3.5 years
  A center-level variable. Exposure to the HKTP is expected to increase the number of Hispanic living kidney donors
number of Hispanic ESRD patients added to the waiting list | Post-intervention exposure up to 3.5 years
  A center-level variable.
number of Hispanic potential donors per potential recipient | Post-intervention exposure up to 3.5 years
  A center-level variable.

OTHER OUTCOMES:
satisfaction with culturally competent care | in year 1-2 and year 4.5
  A center-level variable. The CAHPS survey questionnaire will be used. A mean level of satisfaction will be prospectively comparing routine care with culturally competent care.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa J Gordon, PhD, Principal Investigator — Northwestern University; Juan Carlos J Caicedo, MD, Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - Mayo Clinic Arizon, Phoenix, Arizona
  - University of Colorado Denver, Denver, Colorado
  - Baylor University Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gordon EJ, Lee J, Kang RH, Caicedo JC, Holl JL, Ladner DP, Shumate MD. A complex culturally targeted intervention to reduce Hispanic disparities in living kidney donor transplantation: an effectiveness-implementation hybrid study protocol. BMC Health Serv Res. 2018 May 16;18(1):368. doi: 10.1186/s12913-018-3151-5. PMID 29769080
- [Result] Wang A, Caicedo JC, McNatt G, Abecassis M, Gordon EJ. Financial Feasibility Analysis of a Culturally and Linguistically Competent Hispanic Kidney Transplant Program. Transplantation. 2021 Mar 1;105(3):628-636. doi: 10.1097/TP.0000000000003269. PMID 32282660
- [Result] Gordon EJ, Romo E, Amortegui D, Rodas A, Anderson N, Uriarte J, McNatt G, Caicedo JC, Ladner DP, Shumate M. Implementing culturally competent transplant care and implications for reducing health disparities: A prospective qualitative study. Health Expect. 2020 Dec;23(6):1450-1465. doi: 10.1111/hex.13124. Epub 2020 Oct 9. PMID 33037746
- [Derived] Gordon EJ, Uriarte JJ, Anderson N, Romo E, Caicedo JC, Shumate M. Implementation and modification of an organizational-level intervention: a prospective analysis. Implement Sci Commun. 2022 Jun 3;3(1):59. doi: 10.1186/s43058-022-00296-0. PMID 35659156
- [Derived] Gordon EJ, Lee J, Kang R, Caicedo JC. Impact of having potential living donors on ethnic/racial disparities in access to kidney transplantation. Am J Transplant. 2022 Oct;22(10):2433-2442. doi: 10.1111/ajt.17090. Epub 2022 May 24. PMID 35524363
- [Derived] Gordon EJ, Uriarte JJ, Lee J, Kang R, Shumate M, Ruiz R, Mathur AK, Ladner DP, Caicedo JC. Effectiveness of a culturally competent care intervention in reducing disparities in Hispanic live donor kidney transplantation: A hybrid trial. Am J Transplant. 2022 Feb;22(2):474-488. doi: 10.1111/ajt.16857. Epub 2021 Oct 17. PMID 34559944
- [Derived] Alhalel N, Francone NO, Salazar AM, Primeaux S, Ruiz R, Caicedo JC, Gordon EJ. Patients' perceptions of a culturally targeted Hispanic Kidney Transplant Program: A mixed methods study. Clin Transplant. 2019 Jun;33(6):e13577. doi: 10.1111/ctr.13577. Epub 2019 May 23. PMID 31034642